CLINICAL TRIAL: NCT04796922
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled Study of Parsaclisib Plus Investigator's Choice of Either Rituximab or Obinutuzumab in Participants With Relapsed or Refractory Follicular Lymphoma and Marginal Zone Lymphoma
Brief Title: To Evaluate Efficacy and Safety of Parsaclisib Plus Either Rituximab or Obinutuzumab in R/R Follicular Lymphoma (FL) and Marginal Zone Lymphoma (MZL) (CITADEL-302)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was withdrawn due to a business decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 50465-302
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Follicular Lymphoma ( FL); Marginal Zone Lymphoma (MZL)
Keywords: parsaclisib; Relapsed/Refractory; obinutuzumab; rituximab
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Recurrence | interventions — parsaclisib; Rituximab; obinutuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group A (Experimental): Participants will be administered with parsaclisib in combination with investigator choice of rituximab or obinutuzumab.
  Interventions: Drug: parsaclisib; Drug: rituximab; Drug: obinutuzumab
- Treatment Group B (Placebo Comparator): Participants will be administered with placebo in combination with investigator choice of rituximab or obinutuzumab
  Interventions: Drug: rituximab; Drug: obinutuzumab

INTERVENTIONS:
Drug: parsaclisib — parsaclisib will be administered once daily at 20 mg for 8 weeks followed by 2.5 mg once daily.
  Other Names: INCB050465
  Arms: Treatment Group A
Drug: rituximab — rituximab will be administered intravenously on select days as per protocol.
Drug: obinutuzumab — obinutuzumab will be administered intravenously on select days as per protocol.

SUMMARY:
This is a Phase 3, double-blind, randomized, placebo-controlled, multicenter study of parsaclisib plus investigator's choice of either rituximab or obinutuzumab versus placebo plus investigator's choice of rituximab or obinutuzumab for the treatment of participants with R/R FL or MZL. The Participants will be stratified in a 1:1 randomization ratio by investigator's choice of rituximab or obinutuzumab prior to randomization, time since last antilymphoma therapy (≤ 2, > 2 years), and disease histology (MZL or FL) .

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 years or older (Japan, aged 20 years or older).
* Histologically confirmed Grade 1, 2, or 3a FL or nodal MZL, splenic MZL, or extra nodal MZL
* Prior systemic treatment with at least 1 anti-CD20 mAb (either as monotherapy or in combination as chemoimmunotherapy)
* Documented disease that has relapsed or progressed or was refractory after the most recent prior systemic therapy. Note: Participants must not be refractory to anti-CD20 mAb
* Radiographically (CT, MRI) measurable lymphadenopathy per the Lugano criteria for response assessment (Cheson et al 2014).
* ECOG PS of 0 to 2
* Adequate organ functions including hematopoiesis, liver, and kidney
* Willingness to avoid pregnancy or fathering children

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Known histological transformation from indolent NHL to an aggressive NHL (eg, diffuse large B-cell lymphoma).
* Presence of CNS lymphoma (either primary or secondary) or leptomeningeal disease.
* Prior treatment with PI3K inhibitors.
* Inadequate washout of immunosuppressive therapy, anticancer medications and investigational drugs.
* Significant concurrent, uncontrolled medical condition, including, but not limited to, renal, hepatic, hematological, GI, endocrine, pulmonary, neurological, cerebral, cardiac, infectious, or psychiatric disease.
* Known HIV infection.
* HBV or HCV infection: Participants positive for HBsAg or anti-HBc will be eligible if they are negative for HBV-DNA; these participants must receive prophylactic antiviral therapy. Participants positive for HCV antibody will be eligible if they are negative for HCV-RNA.
* History of other malignancy within 2 years of study entry.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2028-12-20 (Estimated); Study Completion 2032-08-25 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) in R/R FL and MZL participants | 62 months
  Defined as the time from the date of randomization until the first documented disease progression as determined by IRC based on the Lugano criteria for response assessment (Cheson et al 2014) or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) in R/R FL participants | 62 months
  Defined as the time from the date of randomization until the first documented disease progression as determined by IRC based on the Lugano criteria for response assessment (Cheson et al 2014) or death from any cause, whichever occurs first.
Overall Response Rate (ORR) | 62 months
  Defined as the proportion of participants with a CR or PR as determined by IRC based on the Lugano criteria for response assessment (Cheson et al 2014).
Overall Survival (OS) | 10 years
  Defined as the time from the date of randomization until death from any cause.
Progression Free Survival (PFS) in R/R MZL participants | 62 months
  Defined as the time from the date of randomization until the first documented disease progression as determined by IRC based on the Lugano criteria for response assessment (Cheson et al 2014) or death from any cause, whichever occurs first.
Complete Response Rate (CRR) | 62 months
  Defined as the proportion of participants with a CR as determined by IRC based on the Lugano criteria for response assessment (Cheson et al 2014).
Duration of Response (DOR) | 62 months
  Defined as the time from the date of first documented evidence of CR or PR until the first documented disease progression or death from any cause, whichever occurs first, among participants who achieve an objective response as determined by IRC based on the Lugano criteria for response assessment (Cheson et al 2014).
Disease Control Rate (DCR) | 62 months
  Defined as the proportion of participants who achieve best overall response of CR, PR, or SD (Cheson et al 2014) as determined by IRC.
Event Free Survival (EFS) | 62 months
  Defined as the time from the date of randomization to the first documented disease progression as determined by radiographic disease assessment provided by IRC, the initiation of a new antilymphoma therapy, or death from any cause, whichever occurs first.
Time To Next antiLymphoma Therapy (TTNLT) | 62 months
  Defined as the time from the date of randomization to the first documented administration of a new antilymphoma therapy.
Progression-Free Survival on next antilymphoma therapy (PFS2) | 62 months
  Defined as the time from the date of randomization to the first documented disease progression as reported by the investigator after the initiation of a new antilymphoma therapy, death from any cause, or start of a third antilymphoma therapy since randomization in the study, whichever occurs first.
Number of Treatment Emergent Adverse Events (TEAE's) | 62 months
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency